CLINICAL TRIAL: NCT05465278
Title: Clinical Trial to Evaluate the Effect of Alirocumab on the Volume, Architecture and Composition of Atherosclerotic Plaque in Patients With Familial Hypercholesterolemia
Brief Title: Alirocumab and Plaque Burden In Familial Hypercholesterolaemia
Acronym: ARCHITECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Hipercolesterolemia Familiar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARCHITECT
Record Dates: First submitted 2021-07-27; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — alirocumab

STUDY DESIGN:
Intervention Model Description: Low-intervention, open-label, multicenter, phase IV clinical trial to evaluate the effect 18 months after initiation of alirocumab (Praluent®) on the volume, architecture, and composition of the coronary atheroma plaque in subjects with FH and without clinical cardiovascular disease followed in the SAFEHEART registry in optimized and stable treatment with maximum tolerated doses of statins with or without other lipid-lowering treatments under clinical practice conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Alirocumab (Experimental): Every patient enrolled witll receive treatment witl Alirocumab
  Interventions: Drug: Alirocumab

INTERVENTIONS:
Drug: Alirocumab — 18 months treatment with alirocumab

SUMMARY:
Low-level, open-label, multicenter clinical trial to evaluate the effect of alirocumab on the volume, architecture and composition of atherosclerotic plaque in patients with Familial hypercholesterolemia from the SAFEHEART Registry. ARCHITECT study

DETAILED DESCRIPTION:
DISEASE UNDER STUDY Heterozygous familial hypercholesterolemia (FH).

MAIN PURPOSE OF THE TEST The main objective is to evaluate the effect of alirocumab on the burden of coronary atherosclerosis, based on the change in the percentage of volume of atheroma (PVA) by quantifying the atheroma plaque and virtual histology in the entire coronary tree based on the Analysis of coronary CT angiography (CTA) in asymptomatic subjects with FH on optimized and stable treatment with the maximum tolerated doses of statins with or without other lipid-lowering treatments.

MAIN VALUATION VARIABLE The primary endpoint is the change in PVA, throughout the coronary tree, from baseline assessment (before initiation of alirocumab treatment) to 18 months after initiation of alirocumab treatment, based on CTA images analyzed by the QAngio CT software.

DESIGN Low-intervention, open-label, multicenter, phase IV clinical trial to evaluate the effect 18 months after initiation of alirocumab (Praluent®) on the volume, architecture, and composition of the coronary atheroma plaque in subjects with FH and without clinical cardiovascular disease followed in the SAFEHEART registry in optimized and stable treatment with maximum tolerated doses of statins with or without other lipid-lowering treatments under clinical practice conditions.

The study will be carried out in the internal medicine, lipid, endocrinology, and cardiology units of approximately 30 Spanish hospitals.

As it is a low-intervention clinical trial, treatment with alirocumab will be administered according to the terms of the marketing authorization for Praluent®, and the complementary diagnostic and follow-up procedures will entail minimal risk or additional burden for the safety of the patients. subjects, being comparable with that of usual clinical practice.

Patients with FH will be included in whom adequate control of LDL-C levels (LDL-C> 100 mg / dL) is not achieved with the maximum tolerated doses of statins with or without other lipid-lowering agents, in whom the investigator has considered adequate their treatment with alirocumab individually according to their clinical criteria, and based on the indication of this treatment in this patient profile. The study treatment will therefore be the same treatment that the patient would receive even if they did not participate in the study.

The expected duration of the study recruitment period is approximately 6 months. The duration of the study will be 18 months from the inclusion of the last patient.

Once the informed consent of the patients has been obtained, the pertinent evaluations will be carried out to determine the suitability of the patients to participate in the study for a maximum period of 60 days. Once compliance with all the inclusion criteria, and none of the exclusion criteria, has been confirmed, patients will start treatment with alirocumab.

The study follow-up period will be 18 months from the start of treatment. The study follow-up visits will take place at 3 and 12 months (± 30 days), and the final patient visit in the study will take place 18 months (± 30 days) from the start of the study or in case of premature withdrawal. of the patient for reasons other than withdrawal of consent by the patient, loss of follow-up or death. The patients will be followed and treated according to the usual clinical practice during the study period.

The quantification and characterization of coronary atherosclerosis will be evaluated using a coronary CTA. Patients must have availability of an ACT performed in the 3 months prior to the start of the study, and in the event that such evaluation is not available in this period, a coronary CTA will be performed during the selection period. Subsequently, a second THA will be performed 18 months after the start of treatment. The effect of treatment on coronary atherosclerosis will be assessed based on the change in PVA and normalized total atheroma volume (VTA), and the change in the composition and architecture of the coronary wall, by quantifying plaque and Virtual histology in the entire coronary tree measured by coronary CTA, and processed and analyzed using QAngio CT software (Medis medical imaging system, Leiden, the Netherlans).

All the CTAs (baseline and at 18 months) will be analyzed and processed, centrally in the Cardiovascular Imaging Unit of the Hospital Clínico San Carlos (Madrid). During the selection period, the ATC images will be sent through the CRD-e in order to verify that the images obtained meet the technical criteria necessary for them to be properly processed using the QAngio CT software and confirm the presence of a PVA> 30%. so that the patient can be included in the study. 18 months after the start of treatment, the images of the second CTA will be sent through the same procedure as the baseline assessment. The team that analyzes the images using said software to obtain the parameters of the coronary tree will receive the images identified only by a numerical code, so that they will not have access to the personal identifying data of the patient, nor to the clinical data of the patient.

STUDY TREATMENT Patients with FH outside the lipid target (defined by LDL-C levels> 100 mg / dL) will be included in optimized treatment, candidates to receive treatment with alirocumab (Praluent®) 150 mg every 2 weeks subcutaneously, according to the characteristics of the patient. patient with FH and the criteria of the investigator.

As it is a low-intervention clinical trial, the treatment will be administered according to the authorized technical sheet for Praluent® in Spain, and under normal clinical practice conditions.

Participating patients will receive maximized treatment for HF with alirocumab and maximum tolerated doses of statins with or without other lipid-lowering drugs during the study under clinical practice conditions.

Given that it is a study under clinical practice conditions, the study treatment (Praluent®) will be administered following the usual channels of prescription and supply through the hospital pharmacy.

POPULATION UNDER STUDY AND TOTAL NUMBER OF PATIENTS

* Study population: Patients from a subgroup of the SAFEHEART study, adults, of both sexes with a molecular diagnosis of FH, asymptomatic, uncontrolled (defined as LDL-C> 100 mg / dL) with the maximum tolerated doses will be included consecutively. of statins with or without another lipid-lowering treatment, in which it has been decided to start treatment with alirocumab. In addition, all patients must meet all the inclusion criteria and none of the exclusion criteria established in this protocol.
* Total number of patients: The participation of approximately 162 patients distributed in approximately 30 Spanish hospitals is expected.

SCHEDULE AND ESTIMATED DATE OF REALIZATION

The following study schedule is foreseen:

* Presentation of the study to the CEIm: January 2018.
* Approval of the study (CEIm and AEMPS): April 2018
* Inclusion period: May 2018 - October 2018 (6 months).
* Follow-up period: Until April 2020 (18 months after the inclusion of the last patient in the study).
* Closing of the database: September 2020.
* Statistical analysis: November 2020.
* Final report of the study: January 2021. The times described in this calendar may be modified by the administrative deadlines for starting the study.

ELIGIBILITY:
Inclusion Criteria:

* Have voluntarily granted informed consent (preferably in writing or, failing that, orally before independent witnesses of the research team) before carrying out the specific procedures of the trial.
* Patients of both sexes aged between 35 and 65 years.
* Patients with a molecular diagnosis of heterozygous HF included in the Spanish SAFEHEART registry (http://safeheart.colesterolfamiliar.org/).
* Asymptomatic patients.
* Patients without a previous history of clinical cardiovascular events (acute myocardial infarction [AMI], stroke, coronary revascularization, etc.).
* Patients on optimized and stable treatment with maximum tolerated doses of a statin with or without other lipid-lowering therapies, for at least 3 months, with inadequate control, defined by a LDL-C level> 100 mg / dL.
* Availability of a coronary CTA performed in the 3 months prior to the baseline visit. If a coronary CTA is not available, this test will be performed during the selection period.
* ATC of at least 64 cuts performed in a center with sufficient experience (more than 100 ACTs per year).
* Patients with a PVA> 30% in the baseline coronary CTA, performed in the last 3 months before the baseline visit.
* Patients in whom treatment with alirocumab 150 mg / mL is indicated, according to the characteristics of the patient and the Praluent® technical data sheet.

Exclusion Criteria:

* Class> II heart failure according to the functional classification of the NYHA scale (New York Heart Association).
* Heart rate different from normal sinus rhythm (regular HR between 60-100 bpm).
* Previous history of AMI, angina, peripheral arterial thrombosis, stroke or transient ischemic attack (TIA).
* Uncontrolled hypertension defined as a resting systolic blood pressure value> 180 mmHg at the baseline visit.
* Fasting triglyceride levels> 250 mg / dl at baseline visit.
* Type 1 diabetes or insufficiently controlled type 2 diabetes (HbA1> 9%).
* Personal or family history of inherited muscle disorders.
* Known thyroid disease or thyroid replacement therapy.
* Glomerular filtration rate <60 ml / min / 1.73 m2 at baseline visit.
* Elevated ALT and / or AST levels (> 3 times the ULN at the baseline visit).
* Elevated creatinine kinase levels (> 3 times ULN at baseline).
* Patients who have previously received iPCSK9, CETP (cholesterol ester transport protein) inhibitors, mipomersen and / or lomitapide.
* Patients with statin intolerance.
* Active cancer or previous history of cancer.
* Clinically relevant active infection or clinically significant hematologic, renal, metabolic, gastrointestinal, or endocrine dysfunction.
* Availability of a baseline coronary ACT that does not meet the technical requirements for the images to be adequately processed using the QAngio CT software.
* Patient being treated with any investigational drug / product or participating in a clinical trial using an investigational product, with the exception of studies in which the study treatment has been completed more than 6 months ago.
* Pregnant or breast-feeding women, and sexually active women of childbearing potential who are unwilling to use an adequate contraceptive method (such as oral contraceptives, intrauterine device, or barrier method of contraception along with spermicide or surgical sterilization) during the study. Women of childbearing age are defined as those women who have not undergone permanent infertility procedures or who have been amenorrheic for less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change in atherosclerotic plaque burden (%) assessed by coronary computed tomography | 18 months
  change in plaque burden assessed by coronary computed tomography at enrollemnt and at follow-up. Coronary plaque burden and its cgaracteristics will be analysed ant enrollment and at the end of the follow-up

SECONDARY OUTCOMES:
Changue in plaque volume (mm3) assessed by coronary computed tomography | 18 months
  Change in plaque volume assessed by coronary computed tomography at enrollement and at follow up. Coronary plaque volume will be analysed ant enrollment and at the end of the follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion Hipercolesterolemia Familiar, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Perez de Isla L, Diaz-Diaz JL, Romero MJ, Muniz-Grijalvo O, Mediavilla JD, Argueso R, de Andres R, Fuentes F, Sanchez Munoz-Torrero JF, Rubio P, Alvarez-Banos P, Manas D, Suarez Gutierrez L, Saltijeral Cerezo A, Mata P; SAFEHEART Investigators. Characteristics of Coronary Atherosclerosis Related to Plaque Burden Regression During Treatment With Alirocumab: The ARCHITECT Study. Circ Cardiovasc Imaging. 2024 Jan;17(1):e016206. doi: 10.1161/CIRCIMAGING.123.016206. Epub 2024 Jan 11. PMID 38205656
- [Derived] Perez de Isla L, Diaz-Diaz JL, Romero MJ, Muniz-Grijalvo O, Mediavilla JD, Argueso R, Sanchez Munoz-Torrero JF, Rubio P, Alvarez-Banos P, Ponte P, Manas D, Suarez Gutierrez L, Cepeda JM, Casanas M, Fuentes F, Guijarro C, Angel Barba M, Saltijeral Cerezo A, Padro T, Mata P; SAFEHEART Study Group. Alirocumab and Coronary Atherosclerosis in Asymptomatic Patients with Familial Hypercholesterolemia: The ARCHITECT Study. Circulation. 2023 May 9;147(19):1436-1443. doi: 10.1161/CIRCULATIONAHA.122.062557. Epub 2023 Apr 3. PMID 37009731